CLINICAL TRIAL: NCT00575471
Title: A Randomized, Double-Blind, Placebo-Controlled 12-Week Dose-Response Study of Rivoglitazone (CS-011) in Patients With Type 2 Diabetes.
Brief Title: Placebo Controlled Dose-Response Study of Rivoglitazone in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Mr. Yasuhiro Honsho, Daiichi Sankyo Co. Ltd.
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS011-A-J204
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes
Keywords: rivoglitazone HCl; thiazolidinedione; peroxisome proliferator-activated receptor gamma (PPARgamma); diabetes mellitus, type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Carotid Intimal Medial Thickness 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): rivoglitazone HCl 0.5 mg tablets once daily for 12 weeks
  Interventions: Drug: Rivoglitazone HCl
- 2 (Experimental): rivoglitazone HCl 1 mg tablets once daily for 12 weeks
  Interventions: Drug: rivoglitazone HCl
- 3 (Experimental): rivoglitazone HCl 1.5 mg tablets once daily for 12 weeks
  Interventions: Drug: rivoglitazone HCl
- 4 (Placebo Comparator): Matching placebo tablets once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivoglitazone HCl — 0.5 mg tablets once daily for 12 weeks
  Arms: 1
Drug: rivoglitazone HCl — 1.0 mg tablets once daily for 12 weeks
  Arms: 2
Drug: rivoglitazone HCl — 1.5 mg tablets once daily for 12 weeks
  Arms: 3
Drug: Placebo — Matching placebo tablets once daily for 12 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to assess the efficacy response of rivoglitazone HCl on the change in HbA1c after 12 weeks of treatment in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* HbA1c >6.5% and <10%
* FPG >126 mg/dL (7mmol/L) and <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* history of type 1 diabetes
* history of ketoacidosis
* current insulin therapy
* C-peptide <0.5ng/mL
* impaired hepatic function
* CHF or history of CHF (NYHA stage I - IV)
* uncontrolled hypertension

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline for rivoglitazone compared to placebo | 12 weeks

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose from baseline for rivoglitazone HCl compared to placebo | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Fukuoka
  - Osaka
  - Tokyo